CLINICAL TRIAL: NCT02703701
Title: Effects of Provider-at-Triage on Emergency Department Efficiency, Information Delivery and Patient Satisfaction
Brief Title: Role of Provider-at-Triage on ED Efficiency and Quality of Care
Acronym: MD at Triage
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201500586
Record Dates: First submitted 2016-02-23; First posted 2016-03-09 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Patient Satisfaction With Emergency Department Efficiency
Keywords: Patient Satisfaction; Emergency Department efficiency
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Usual Care: Group enrolled during normal emergency department operating procedures (without a physician present at triage).
  Interventions: Other: Usual Care
- Physician at Triage: Group enrolled while a physician is present at triage.
  Interventions: Behavioral: Physician at triage

INTERVENTIONS:
Behavioral: Physician at triage — A physician embedded at triage
  Groups: Physician at Triage
Other: Usual Care — No physician at triage
  Groups: Usual Care

SUMMARY:
The United States spends over $8,000 per capita annually on health care and its health care system is more expensive than other developed countries. Even with high per capita costs and a high proportion of physician specialists, the US lags in health care performance from patients' perspectives.

The hospital emergency department (ED) is often the portal of entry for patients seeking health care services and is therefore an ideal setting for initiatives to improve efficiency of care delivery and patient satisfaction. Reduction in wait times, enhanced information delivery and ED staff service quality all have a positive influence on patient perception of health care quality and satisfaction.

Prior studies have attempted to increase patient satisfaction by improving staff communication and courtesy, implementing a patient satisfaction team in triage, and delivering information to patients in a timely manner. Another strategy to increase the efficiency of ED operations is adding a physician to triage to perform brief medical screenings and initiate necessary patient testing and treatment. This contrasts to usual practice in which physicians evaluate patients only following registration and nurse assessment of illness or injury severity.

DETAILED DESCRIPTION:
This study will assess the impact of early patient assessment by a physician at Emergency Department (ED) triage on patient perception of information delivery, overall patient satisfaction and ED efficiency. ED efficiency will be assessed by ED length of patient stay, ED left-without-being-seen and ED left during treatment rates.

Participants who decide to take part in this study, will be asked questions by research staff, who will document responses on a secure iPAD device. The survey will ask participants how they feel about their health condition, the emergency department wait, the care they received in the emergency department and how satisfied the participant was with the care received.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to participate in the study if they are:

* English speaking
* Without hemodynamic or respiratory compromise
* Do not have a nurse-assigned triage severity score of Emergency Severity Index 1 (most severe illness or injury score).

Exclusion Criteria:

Participants will be excluded if they are:

* Unwilling or unable to sign an informed consent
* In police custody
* Too ill to participate in study.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals receiving care from the Emergency Department between 10am-3pm on days a physician is (Monday-Wednesday) and is not (Thursday-Sunday) assigned to triage.
Sampling Method: Non-Probability Sample
Enrollment: 439 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | 60 minutes after Emergency Department triage
  Patient Satisfaction Score- brief survey measured on a Likert Scale
  * 1= Never
  * 2= Sometimes
  * 3= Usually
  * 4= Always
  * 5= Not applicable - I did not see a doctor today

SECONDARY OUTCOMES:
Emergency Department efficiency | 24 hours after ED triage in minutes
  Impact of physician at triage on ED length of stay rates
Left without being seen rate | 12 hours after ED triage in minutes
  Impact of physician at triage on left without being seen rate

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Allen, MD, Principal Investigator — Univeristy of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No